CLINICAL TRIAL: NCT06118749
Title: Leishmania Antigen Rapid Diagnostic Test Proof-of-Concept and Validation Study
Status: Terminated | Type: Observational
Why Stopped: Desk review conducted on study documentation revealing certain inconsistencies leading to the recommendation to halt the study.
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NT015
Record Dates: First submitted 2023-05-10; First posted 2023-11-07 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Visceral Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Antigen detection Rapid Diagnostic Test prototype — The study will focus on the usability and diagnostic performance of the RDT in blood and/or urine from patients with visceral leishmaniasis.

SUMMARY:
Visceral leishmaniasis (VL) or kala azar is a neglected tropical disease(NTD) caused by protozoan parasites of the Leishmania donovani complex that are transmitted by phlebotomine sand flies. An estimated 50,000 - 90,000 new cases occur worldwide annually. It is characterized by fever, weight loss, enlargement of the spleen and liver, and anaemia, and it can be fatal in more than 95% of cases without treatment. The Horn of Africa accounts for the largest number of VL cases worldwide, and communities living in remote, resource-limited settings are at greatest risk of infection. Therefore, early and accurate diagnosis of VL in health facilities is essential. VL is fatal if it is not adequately treated. The drugs currently used to treat VL can have severe side effects and the clinical presentation of VL is not sufficiently specific to guide treatment. Highly accurate (both sensitive and specific), cheap and simple rapid diagnostic tests (RDTs) are therefore crucial for case-management of VL. Early case detection followed by adequate treatment is also central to control of VL.

In Kenya, Visceral leishmaniasis is diagnosed by the rK39 RDT based on detection of host antibody to a 39-aminoacid-repeat recombinant leishmanial antigen in clinically suspected cases. Because this test has a suboptimal sensitivity of around 85%, other additional diagnostic tests are often necessary. These include the direct agglutination test (DAT) based on agglutination of whole parasite antigen by parasite specific host antibodies and microscopy detection of amastigotes in stained smears from lymph node punctures, bone marrow or spleen aspirates currently the gold standard for confirmatory diagnosis.

While the use of rK39 RDT and DAT has been on the increase, the tests cannot distinguish active from past infections as they are based on detection of antileishmania antibodies which are present in both active and past infections. Furthermore, DAT requires some laboratory skills and overnight incubations before obtaining the results and the rK39 has low sensitivity when used in Eastern Africa. There have therefore been efforts to develop an antigen detection based test that is based on minimally invasive specimen collection such as blood or urine.

To this end, a collaboration between KEMRI, DNDi, FIND and the University of York under the Next generation diagnostics and oral treatment for visceral leishmaniasis in Eastern Africa: transforming patient care through innovation (VL-INNO) EDCTP project, aims to develop an antigen based diagnostic test based on parasite biomarkers in urine and blood from VL patients. In this project, a proteomics approach will be used to identify candidate Leishmania antigens that are found in the blood and urine of confirmed visceral leishmaniasis. The University of York will undertake proteomics analyses of the specimens using highly sensitive Liquid Chromatograph Triple Quadrupole Mass Spectrometer (LCMS/MS) to explore antigen diversity in defined archived clinical samples (blood, urine) from VL patients before and after treatment. Based on yield, stability and immunogenicity of the antigens, monoclonal antibodies (mAb) will be production for subsequent development of a lateral flow rapid diagnostic test(RDT) prototype that can detect leishmania antigens in blood and/or urine of VL patients.

With these activities initiated using samples previously collected from VL patients in Kenya, this current protocol seeks to collect samples (blood and urine) from two VL treatment centres namely Chemolingot Sub-county hospital in Baringo County and Kacheliba Sub-county, West Pokot, to be used in the evaluation of the RDT prototype. We will analyze samples from VL patients collected before and at the end of treatment, to determine the sensitivity of the test and how parasite antigen abundance in urine and blood changes as a consequence of clinical cure. Samples from healthy endemic controls will be used to determine the specificity of the test.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if ALL of the following criteria are met:

* Patient with a confirmed diagnosis of VL based on the VL diagnostic algorithm as in the national guidelines, either before treatment or after treatment completion OR healthy individuals with no clinical signs compatible with VL.
* Participant ≥ 4 years old.
* Participant from whom written informed consent can be obtained or signed by parent or legal guardian if patient is under 18 years of age. In the case of minors, assent from the children (13-17 years old) will be obtained.
* Clinical samples required for the study (peripheral blood and urine) can be obtained.

Exclusion Criteria:

Participants cannot be included in the study if ANY of the following criteria apply:

* Patients < 4 years old.
* Patients from which, for any reason, none of the sample needed (urine or blood) can be taken.

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a primary diagnosis of VL, VL patients that are ready for discharge after treatment completion, and healthy individuals accompanying patients, will be consented and recruited at the VL treatment centres in Kacheliba and Chemolingot Sub-county hospitals in West Pokot and Baringo counties.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 18 months
  The diagnostic accuracy of newly developed RDT will be evaluated to give specificity, sensitivity values

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No